CLINICAL TRIAL: NCT01061138
Title: A Multi-Center Clinical Study to Acquire Xpress Digital Mammography System Images for Computer Aided Detection Development
Brief Title: Xpress Digital Mammography System Images for Computer Aided Detection Development
Status: Completed | Type: Observational
Sponsor: Konica Minolta Medical Imaging, USA (Industry)
Responsible Party: Sponsor
Other Study IDs: #03
Record Dates: First submitted 2010-02-01; First posted 2010-02-02 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Breast Cancer
Keywords: breast cancer; screening mammograms; breast biopsy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Screening Patients: Female patients scheduled for routine annual screening mammograms
- Biopsy Patients: Female patients scheduled for routine breast biopsy procedures

SUMMARY:
The primary objective of this study is to acquire digital mammography images produced by the Xpress Digital Mammography System in order to develop Computer Aided Detection software and systems.

DETAILED DESCRIPTION:
The proposed study is an image acquisition study of mammograms produced by the investigational digital system. Women who meet the selection criteria and who agree to participate in the study will be imaged with the Xpress Digital Mammography System at the clinical sites. These images will be provided to CAD development companies to conduct their own development and testing. The CAD development companies will be responsible for submitting their results to the FDA for marketing approval of their CAD systems.

Patients will be drawn primarily from those women scheduled for breast biopsy since this population has an enhanced probability of cancer. The intent is to enroll patients until at least 107 women with biopsy proven cancers, and at least 330 women who have negative mammograms are enrolled. All cancers found will be used in the study. It is anticipated that approximately 720 patients undergoing diagnostic mammography will need to be enrolled to yield 107 proven cancer cases. In addition, approximately 330 cases will be drawn from a screening population. The negative status of the screening cases will be established by selecting only cases classified as BIRADS 1 or 2, and have a negative mammogram at one year follow-up. All images collected will be utilized to develop and test the CAD systems, and may be used for further product development.

ELIGIBILITY:
Inclusion Criteria

Cases selected for the study must meet all of the following criteria:

* Female
* Scheduled for a routine screening mammography or routine breast biopsy for non-palpable findings
* Any ethnic origin

Exclusion Criteria

Patients meeting any of the following criteria will be excluded from the study:

* Any contraindication to mammography
* Pregnant or suspicion of being pregnant, or nursing
* Patients with palpable lesions
* Patients with internal breast markers in the region of interest
* Breast implants, without displaced views
* Significant recent breast trauma/acute mastitis
* Patient has previously undergone an excisional breast biopsy
* Patients with a history of breast cancer
* Unable or unwilling to give consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: To achieve the goal of 107 cases with biopsy-proven cancer, it is expected that approximatley 720 patients undergoing breast biopsy will need to be enrolled in the study. In addition, we will enroll up to 330 patients from a screening population.
Sampling Method: Non-Probability Sample
Enrollment: 597 (Actual)
Dates: Start 2010-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Etta Pisano, MD, Principal Investigator — Medical University of South Carolina
Locations (5):
- United States (5):
  - Waterbury Hospital, Waterbury, Connecticut
  - Jackson Memorial Hospital, Miami, Florida
  - University of Iowa, Iowa City, Iowa
  - Greenville Hospital Systems, Greenville, South Carolina
  - University of Texas San Antonio, San Antonio, Texas